CLINICAL TRIAL: NCT05925127
Title: A Phase 2/3, Randomized, Double-Blind Study to Evaluate the Safety and Immunogenicity of Different Booster Dose Levels of Monovalent SARS-CoV-2 rS Vaccines in Adults ≥ 50 Years Previously Vaccinated With COVID-19 mRNA Vaccines
Brief Title: Phase 2/3 Heterologous Boosting Study With Different Dose Levels of Monovalent SARS-CoV-2 rS Vaccines
Acronym: COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2019nCoV-205
Record Dates: First submitted 2023-06-27; First posted 2023-06-29 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Group-A Monovalent NVX-CoV2373 (5 μg) (Experimental): The Monovalent NVX-CoV2601 of 5 μg of antigen with 50 μg of Matrix-M adjuvant
  Interventions: Biological: NVX-CoV2373 (5μg)
- Group-B Monovalent NVX-CoV2601 (5 μg) (Experimental): Monovalent NVX-CoV2601 (5 μg of antigen with 50 μg of Matrix-M adjuvant)
  Interventions: Biological: NVX-CoV2601 (5μg)
- Group-C Monovalent NVX-CoV2601 (5 μg) (Experimental): Monovalent NVX-CoV2601 (5 μg of antigen with 75 μg of Matrix-M adjuvant)
  Interventions: Biological: NVX-CoV2601(5μg)
- Group-D Monovalent NVX-CoV2601 (35 μg) (Experimental): Monovalent NVX-CoV2373 (35 μg of antigen with 50 μg of Matrix-M adjuvant)
  Interventions: Biological: NVX-CoV2601 (35μg)
- Group-E Monovalent NVX-CoV2601(35) (Experimental): Monovalent NVX-CoV2601 (35 μg of each antigen with a 75 μg of Matrix-M adjuvant)
  Interventions: Biological: NVX-CoV2601(35μg)
- Group-F Monovalent NVX-CoV2601 (50 μg) (Experimental): Monovalent NVX-CoV2601 (50 μg of each antigen with a 100 μg of Matrix-M adjuvant)
  Interventions: Biological: NVX-CoV2601(50μg)
- Group-G Bivalent XBB.1.5 (Experimental): Bivalent XBB.1.5 Omicron subvariant/prototype COVID-19 licensed mRNA vaccine
  Interventions: Biological: Bivalent BA.4/5

INTERVENTIONS:
Biological: NVX-CoV2373 (5μg) — Coformulated prototype SARS-CoV-2 rS vaccine with Matrix-M adjuvant: supplied as a solution for preparation for injection, at a concentration of 10 μg/mL and 100 μg adjuvant per mL, respectively
  Arms: Group-A Monovalent NVX-CoV2373 (5 μg)
Biological: NVX-CoV2601 (5μg) — The vaccination regimen will comprise one IM injection on Day 0 at a dose of 5 µg of antigen with 50 µg Matrix-M adjuvant.
  Other Names: Omicron XBB.1.5
  Arms: Group-B Monovalent NVX-CoV2601 (5 μg)
Biological: NVX-CoV2601(5μg) — The vaccination regimen will comprise one IM injection on Day 0 at a dose of 5 µg of antigen with 75 µg Matrix-M adjuvant.
  Other Names: Omicron XBB.1.5
  Arms: Group-C Monovalent NVX-CoV2601 (5 μg)
Biological: NVX-CoV2601 (35μg) — The vaccination regimen will comprise one IM injection on Day 0 at a dose of 35 µg of antigen with 50 µg Matrix-M adjuvant.
  Other Names: Omicron XBB.1.5
  Arms: Group-D Monovalent NVX-CoV2601 (35 μg)
Biological: NVX-CoV2601(35μg) — The vaccination regimen will comprise one IM injection on Day 0 at a dose of 35 µg of antigen with 75 µg Matrix-M adjuvant.
  Other Names: Omicron XBB.1.5
  Arms: Group-E Monovalent NVX-CoV2601(35)
Biological: NVX-CoV2601(50μg) — The vaccination regimen will comprise one IM injection on Day 0 at a dose of 50 µg of antigen with 100 µg Matrix-M adjuvant
  Other Names: Omicron XBB.1.5
  Arms: Group-F Monovalent NVX-CoV2601 (50 μg)
Biological: Bivalent BA.4/5 — The bivalent BA.4/5 (or recommended mRNA vaccine at the time of the conduct of this study) Omicron subvariant/prototype licensed mRNA vaccine will be procured and stored per the manufacturer's instructions. For this vaccine group, treatment will be administered open label as a single IM injection
  Other Names: Omicron Subvariant/Prototype Licensed mRNA Vaccine
  Arms: Group-G Bivalent XBB.1.5

SUMMARY:
This is a Phase 2/3, randomized, double-blind study to evaluate the safety and immunogenicity of different booster dose levels of the monovalent severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) recombinant (r) spike (S) protein nanoparticle (SARS-CoV-2 rS) vaccines with Matrix-M™ adjuvant (NVX-CoV2373 [prototype Wuhan vaccine with Matrix-M adjuvant] or NVX-CoV2601 [Omicron XBB.1.5 subvariant vaccine with Matrix-M adjuvant]).

DETAILED DESCRIPTION:
The ongoing COVID-19 pandemic has reached a stage where it is necessary to stablish the framework for periodic national vaccination campaigns.The present study aims to investigate the safety and immunogenicity of different booster dose levels of monovalent and bivalent vaccines in adults ≥ 50 years of age who have already been immunized with ≥ 3 doses of a COVID-19 prototype or bivalent licensed mRNA vaccine. The Boosters of investigational products will be administered ≥ 90 days after the participants received their third dose of a COVID-19 prototype or bivalent licensed mRNA vaccine.

Approximately 1,980 participants ≥ 50 years of age who have received a regimen of ≥ 3 doses of a coronavirus disease 2019(COVID-19) vaccine (the last vaccine could have been a bivalent licensed mRNA vaccine) will be included in this study. The last COVID-19 vaccine dose should have been administered ≥ 90 days prior to Day 0.

Approximately 1,800 participants will be randomly assigned in a 1:2:2:2:2:1 ratio to receive NVX-CoV2373 or NVC-CoV2601 in a double-blinded fashion into 1 of 6 monovalent vaccine groups (vaccine groups A to G). Following completion of enrollment into the 6 monovalent vaccine groups, 180 participants will be enrolled in vaccine group G to receive a bivalent licensed mRNA vaccine in an open-label fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 50 years of age at screening.
2. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
3. Female participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea ≥ 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from ≥ 28 days prior to enrollment and through the end of the study.
4. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to the initial study vaccination.
5. Agrees to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study.
6. Have previously received ≥ 3 doses of a COVID-19 prototype or bivalent licensed mRNAvaccine with the last dose having been given ≥ 90 days previously prior to first study booster.

Exclusion Criteria:

1. Received COVID-19 vaccines other than a COVID-19 prototype or bivalent licensed mRNA vaccine in the past, inclusive of clinical trial COVID-19 vaccines.
2. Participation in research involving receipt of investigational products (drug/biologic/device) within 90 days prior to study vaccination.
3. Received influenza vaccination within 14 days prior to first study vaccination, or any other vaccine within 30 days prior to first study vaccination.
4. Any known allergies to products contained in the investigational product. 5. Any history of anaphylaxis to any prior vaccine.

6. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) requiring ongoing immunomodulatory therapy.

7. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to study vaccination. NOTE: An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical or intranasal glucocorticoids is permitted. Topical tacrolimus and ocular cyclosporin are permitted. Use of inhaled glucocorticoids is prohibited.

8. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to study vaccination, except for rabies immunoglobulin which may be given if medically indicated.

9. Active cancer (malignancy) on therapy within 3 years prior to study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).

10. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study.

11. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to the study vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.

12. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).

13. Study team member or immediate family member of any study team member (inclusive of Sponsor, contract research organization (CRO), and study site personnel involved in the conduct or planning of the study).

14. Participants with a history of myocarditis or pericarditis.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 994 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-Neutralizing antibody expressed as geometric mean titer ratio[GMTR ]against the Omicron subvariant XBB.1.5 | Day 28
  Neutralizing antibody To determine if the combination of antigen and adjuvant levels of NVX-CoV2601 GMTR against the Omicron subvariant XBB.1.5 superior(LB of the 95% CI for GMTR > 1.0) to that elicited by NVX-CoV2373
Immunogenicity index-Neutralizing antibody expressed as seroresponse rates (SRRs)against the Omicron subvariant XBB.1.5 | Day 28
  Neutralizing antibody SRR against the Omicron XBB.1.5 subvariant elicited by NVXCoV2601 is non-inferior (NI)to the SRR elicited by NVX-CoV2373in participants ≥ 50 years of age previously vaccinated with ≥ 3 doses of a COVID-19 prototype or bivalent licensed mRNA vaccine.

SECONDARY OUTCOMES:
Neutralizing antibody expressed as geometric mean titer ratio[GMTR ]against the Omicron subvariant XBB.1.5 | Day 28
  Neutralizing antibody (GMTR) at relevant time points Days 28 to 180 from baseline (Day 0) and analyzed by dose (5, 10, and 25 µg)
Immunogenicity index- IgG antibody Anti-S expressed as geometric mean Elisa units GMEUs (EU/mL) | Day 0 to 180
  Immunoglobulin G (IgG) antibody Anti-S expressed as geometric mean Elisa units GMEUs (EU/mL) at relevant time points (Days 0 to 180) and analyzed by dose (5, 10, and 25 µg)
Immunogenicity index- Neutralizing antibody titers of post-booster by baseline anti-SARS-CoV-2 NP | Day-28
  Neutralizing antibody titers of post-booster by baseline anti-SARS-CoV-2 NP status day-28
Immunogenicity index- Serum IgG levels to SARS-CoV-2 S protein at Day 28 of post-booster | Day-28
  Serum IgG levels to SARS-CoV-2 S protein at Day 28 post-booster by baseline anti-SARS-CoV-2 NP status.
Safety Index-Incidence, duration, and severity of solicited local and systemic AEs expressed as GMT | 7 days
  Incidence, duration, and severity of solicited local and systemic AEs for 7 days following vaccination.
Safety Index -Incidence and relationship of Medically Attended Adverse Event(s) (MAAEs), Adverse event(s) of Special Interest (AESIs), and Serious Adverse Event(s) (SAEs) | Day 0 to 180
  Incidence and relationship of Medically Attended Adverse Event(s) (MAAEs), Adverse event(s) of Special Interest (AESIs), and Serious Adverse Event(s) (SAEs) [ Time Frame: Day 0 to Day 180 ] Incidence and relationship of MAAEs, AESIs (predefined list), and SAEs throughout the study
Safety Index -Incidence, Severity, and relationship of unsolicitated Adverse Event(s) Through 28 days after vaccination by vaccine group p(vaccine groups A to G). | Day 0 to 180
  Incidence, Severity, and relationship of unsolicitated Adverse Event(s) Through 28 days after vaccination by vaccine group p(vaccine groups A to G).s the overall safety of single-dose regimens containing NVX-CoV2601, NVX-CoV2373, or mRNA vaccine by vaccine group in participants ≥ 50 years of age previously vaccinated with ≥ 3 doses of a COVID-19 prototype or bivalentlicensed mRNA vaccine.
Human angiotensin-converting enzyme 2 (hACE2) receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses expressed as GMTs | Day 0 to 180
  hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses at relevant time points (Days 0, 28, and 180) and analyzed by dose (5, 10, and 25 µg)
hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses expressed as GMFR | Day 0 to 180
  hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses at relevant time points (Days 0, 28, and 180) and analyzed by dose (5, 10, and 25 µg).
hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins expressed as SRR | Day 0 to 180
  hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins at relevant time points (Days 0, 28, and 180)and analyzed by previous vaccine combination received. Derived/calculated endpoints based on these data will include SRRs.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax
Locations (49):
- United States (49):
  - ARS-Birmingham CRU, Birmingham, Alabama
  - Tucson Neuroscience Research, Tucson, Arizona
  - Velocity Clinical Research, Banning, Banning, California
  - Velocity Clinical Research, Chula Vista, Chula Vista, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis - San Diego, San Diego, California
  - WR-MCCR, San Diego, California
  - Deland CRU, DeLand, Florida
  - Health Awareness, Jupiter, Florida
  - Wr-Msra, Llc, Lake City, Florida
  - Professional Urgent Care Services, Largo, Florida
  - Research Institute of South Florida, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Headlands Research Orlando LLC, Orlando, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - TrueBlue Clinical Research, Tampa, Florida
  - Neurostudies CRU, Decatur, Georgia
  - Velocity Clinical Research, Savannah, Georgia
  - CRA Headlands LLC, Stockbridge, Georgia
  - Velocity Clinical Research, Meridian, Idaho
  - Velocity Clinical Research, Sioux City, Iowa
  - Velocity Clinical Research, Baton Rouge, Louisiana
  - Velocity Clinical Research - Covington, Covington, Louisiana
  - Velocity Clinical Research, Metairie, Metairie, Louisiana
  - Activmed Practices and Research, LLC, Methuen, Massachusetts
  - Velocity Clinical Research, Gulfport, Gulfport, Mississippi
  - Velocity Clinical Research, Grand Island, Nebraska
  - Velocity Clinical Research, Norfolk, Nebraska
  - Velocity Clinical Research, Omaha, Nebraska
  - Activmed Practices and Research, LLC, Portsmouth, New Hampshire
  - Velocity Clinical Research, Binghamton, New York
  - Hypercore (Lucas Research), New Bern, North Carolina
  - M3 Wake Research Inc, Raleigh, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Javara Inc./Wake Forest Health Network, LLC, Winston-Salem, North Carolina
  - Velocity Clinical Research, Cincinnati, Ohio
  - Tekton Research, Edmond, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Grants Pass, Grants Pass, Oregon
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Velocity Clinical Research, Gaffney, Gaffney, South Carolina
  - Coastal Carolina Research Center an ALCANZA Clinical Research company, North Charleston, South Carolina
  - Central Texas Clinical Research, LLC, Austin, Texas
  - Research Your Health, Plano, Texas
  - Benchmark Research, San Angelo, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Health Research of Hampton Roads, Inc, Newport News, Virginia
  - Clinical Research Partners, Richmond, Virginia